CLINICAL TRIAL: NCT00706329
Title: Study of Minimally Invasive Closure of Umbilical Hernias
Brief Title: Minimally Invasive Closure of Umbilical Hernias
Acronym: MIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated prematurely by the IRB due to data integrity and protocol compliance issues
Sponsor: South Shore Hospital (Other)
Collaborators: Q-Med Scandinavia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSH ID 07-003; NCT00839618 (obsolete NCT alias)
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Umbilical Hernia
Keywords: Minimally invasive surgery; Umbilical hernia; Infant
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deflux (Experimental): Treatment with Deflux.
  Interventions: Device: Deflux

INTERVENTIONS:
Device: Deflux — Patients undergo surgery using Deflux to correct umbilical hernia

SUMMARY:
The purpose of the study is to test the use of "Deflux" injections in a minimally invasive closure of umbilical (belly button) hernias in infants between birth and five years. The study is designed to demonstrate that the use of this device can safely and effectively close an umbilical hernia.

DETAILED DESCRIPTION:
All patients will undergo general anesthesia for their primary procedure, i.e. inguinal hernia repair. Once under general anesthesia, the abdomen will be prepped and draped in the usual sterile surgical fashion. The edge of the umbilical hernia defect will be palpated and in case there are any contents of the hernia present, they will be pushed into the abdominal cavity. Adequate relaxation, again, will be assured. A 24 gauge needle will be used to inject 1cc of Deflux ("Study Product") into each quadrant at the junction between the preperitoneal space and the inner palpable rim of the fascial defect. The surgeon's index finger stays in the center of the hernia defect, protecting the hernia sac contents from re-herniating. Closure of the umbilical defect will be confirmed by palpation immediately after injection. A sterile wound dressing will be applied and the primary surgical procedure will be performed afterwards.

Definition of Primary and Secondary Outcomes/Endpoints:

The endpoint of this study is closure of the umbilical hernia.

Data Collection Methods, Assessments, and Schedule (what assessments performed, how often): A data collection file is started at the time of enrollment in the study. Data collection includes patient age, gender, and weight at the time of operation, inner diameter of the umbilical hernia defect at the time of operation, description of the immediate postoperative results and follow-up exams at two weeks, one month, and six months.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-5 years
* Umbilical hernia>1cm. diameter.
* Undergoing either a general surgical or urologic procedure under general anesthesia other than umbilical hernia repair.
* No previous umbilical hernia repair.

Exclusion Criteria:

* Over 5 years
* No umbilical hernia
* No other surgery required
* Previous umbilical hernia repair

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil R. Feins, M.D., Principal Investigator — Children's Hospital Boston and South Shore Hospital
Locations (1):
- Children's Hospital Boston and South Shore Hospital, South Weymouth, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: physician office
Pre-assignment Details: 59 medical records were screened; 25 were eligible and received Deflux
Period: Overall Study
Arm/Group | Deflux
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated prematurely by the IRB due to data integrity and compliance concerns.
Arm/Group | Deflux
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Close Belly Button or Umbilical Hernia
Description: The study was terminated prematurely by the IRB. Results are not shared due to data integrity concerns. These concerns are outlined in an FDA warning letter.
Time Frame: After surgery, subjects will be followed at intervals of one month and six months from date of surgery.
Arm/Group | Close Belly Button or Umbilical Hernia
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The study was terminated prematurely by the IRB due to data integrity and compliance concerns.
Arm/Group | Deflux
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the IRB due to data integrity and compliance concerns. Results are not shared due to data integrity concerns. These concerns are outlined in an FDA warning letter.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No